CLINICAL TRIAL: NCT06144814
Title: A Comparison of Hyaluronic Acid and Estradiol Treatment in Vulvovaginal Atrophy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koru Health Groups (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KoruHealth
Record Dates: First submitted 2023-11-14; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Vulvovaginal Atrophy
Keywords: vulvovaginal atrophy; Hyaluronic acid; estradiol

STUDY DESIGN:
Intervention Model Description: The objective of this randomized controlled trial was to compare the effect of Hyaluronic acid and Estradiol and to determine the effect on VHI. Secondary objective was to investigate the effect of VVA/GSM on symptoms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyaluronic acid (Experimental): The objective of this randomized controlled trial was to compare the effect of Hyaluronic acid and Estradiol and to determine the effect on VHI.
  Interventions: Drug: Hyaluronic acid vaginal gel
- Estradiol (Active Comparator): Secondary objective was to investigate the effect of Hyaluronic acid to VVA/GSM on symptoms.
  Interventions: Drug: Estrogen vaginal use form

INTERVENTIONS:
Drug: Hyaluronic acid vaginal gel — . Group II received 5 mg of vaginal hyaluronic acid every day for 14 days, then 2 days a week for the next 2 weeks. Hyaluronic acid gel for vaginal use was supplied by ORTHOGEN®. The treatment period lasted 1 month in both groups.
  Arms: Hyaluronic acid
Drug: Estrogen vaginal use form — Group I received 25 µg vaginal estrodiol (Vagifem®). 1 tablet a day for two weeks, then 2 times a week for the next 2 weeks.
  Arms: Estradiol

SUMMARY:
The goal of this observational study isto compare the effect hyaluronic acid and estradiol in vulvo-vaginal atrophy.Hyaluronic acid and Estrogen were equally effective in vaginal treatment. Hyaluronic acid may be preferred for patients in whom hormonal therapy is contraindicated or who wish to receive non-hormonal therapy.

DETAILED DESCRIPTION:
This randomized, controlled, monocentric, prospective, comparative (before/after) study was conducted at Koru Ankara Hospital between April 2023 and September 2023. Patients were randomized into 2 groups. A total of 300 patients, 150 in each group, were included in the study. Informed written consent was obtained from the volunteers who willingly participated in the study. Group I received 25 µg vaginal estrodiol (Vagifem®). 1 tablet a day for two weeks, then 2 times a week for the next 2 weeks. Group II received 5 mg of vaginal hyaluronic acid every day for 14 days, then 2 days a week for the next 2 weeks. Hyaluronic acid gel for vaginal use was supplied by ORTHOGEN®. The treatment period lasted 1 month in both groups.

Before receiving treatment, patients who consented to participate in the study were examined by a Gynecologist, and Vaginal Health Index (VHI)12 score was determined. After the end of the treatment period, the patients were re-evaluated by the same physician, and the VHI score was obtained again. The VHI is the most common score based on vaginal elasticity, secretions, pH, presence of petechiae on the epithelial mucosa, and hydration assessment. The score can range from 5 to 25, and <15 is considered an atrophic vagina index.

Vaginal pH was measured by placing pH paper on the anterior wall of the vagina. A value >5 pH was defined as decreased estrogen activity13. The effect on the primary outcome VHI index was investigated.

ELIGIBILITY:
Inclusion Criteria:

- age over 40 years, FSH value above 25 pg/ml, LH value above 20 pg/ml, E2 value below 15 pg/ml, endometrial thickness of 5 mm or less, and absence of menstruation for 12 months.

Exclusion Criteria:

* patients receiving Hormone Replacement Therapy (HRT), genital organ malignancy, breast cancer, patients with vaginal bleeding of unknown cause, history of thrombophlebitis and thromboembolism, thrombophilia, acute or chronic cardiovascular diseases, estrogen and hyaluronic acid allergy, vaginal infection, acute or chronic cardiovascular diseases, and liver diseases. Patients eligible to participate in the study were required to report at least one of the following symptoms: vaginal dryness, burning or irritation, lack of lubrication during intercourse, sexual discomfort or pain during intercourse, dysuria, or recurrent urinary tract infection.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female only
Enrollment: 300 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
A comparison of hyaluronic acid and estradiol treatment in vulvovaginal atrophy. | 1 month
  Before receiving treatment, patients who consented to participate in the study were examined by a Gynecologist, and Vaginal Health Index (VHI) score was determined. After the end of the treatment period, the patients were re-evaluated by the same physician, and the VHI score was obtained again. The VHI is the most common score based on vaginal elasticity, secretions, pH, presence of petechiae on the epithelial mucosa, and hydration assessment. The score can range from 5 to 25, and <15 is considered an atrophic vagina index.

SECONDARY OUTCOMES:
A comparison of hyaluronic acid and estradiol treatment in vulvovaginal atrophy. | 1 month
  Vaginal pH was measured by placing pH paper on the anterior wall of the vagina. A value >5 pH was defined as decreased estrogen activity. The effect on the primary outcome VHI index was investigated

CONTACTS AND LOCATIONS:
Locations (1):
- Turkey, Ankara, Çankaya, Turkey (Türkiye)